CLINICAL TRIAL: NCT06609642
Title: Digital Art and Artificial Intelligence : Encouraging the Discovery of the Senses Via the Impressionist Painters for the Well-being of Adults - Qualitative Study
Brief Title: Digital Art and Artificial Intelligence
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Olivier Beauchet (Other Government)
Collaborators: Centre integre universitaire de sante et de services sociaux du Centre-Sud-de-l'Île-de-Montréal (Other Government)
Responsible Party: Sponsor-Investigator, Olivier Beauchet, MD PhD, Centre integre universitaire de sante et de services sociaux du Centre-Sud-de-l'Île-de-Montréal
Organization: Centre integre universitaire de sante et de services sociaux du Centre-Sud-de-l'Île-de-Montréal (Other Government)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2025-2244
Record Dates: First submitted 2024-09-18; First posted 2024-09-24 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Adults

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Young adults (Experimental): Male and female, aged 18 to 35 years
  Interventions: Behavioral: Art application
- Old adults (Experimental): Male and female, aged 60 years and more
  Interventions: Behavioral: Art application

INTERVENTIONS:
Behavioral: Art application — First, participants will complete questionnaires that will provide us with their socio-demographic information, their level of knowledge in visual arts and music, as well as their level of eco-anxiety.
  Second, participants will use the application on a touchscreen tablet:
  1. A member of the research team will give a brief explanation of the application.
  2. The participant will use the application on the touchscreen tablet.
  3. A member of the research team will be present in the room during the test as an observer.
  Third, the participant will answer questions from a member of the research team: impressions of the tool, digital skills and abilities, enablers and barriers to the use of the tool, expectations, needs, and interests in the application.

SUMMARY:
The study aims at examining the impact of an immersive and interactive digital application (App) that uses impressionist artworks to promote the mental well-being of both young and older adults. The goal is to study the usability and accessibility of this App, particularly for older adults, who may have sensory impairments and lower digital literacy compared to younger adults.

The study is based on the hypothesis that the App, which allows interaction with paintings by Claude Monet and Helen McNicoll, can trigger positive emotions, thereby improving users' well-being. The App uses artificial intelligence to create extensions of the paintings and music based on the sonification of electrophysiological signals captured from plants.

The study seeks to answer four research questions:

1. The usage behaviors of young and older adults with the App.
2. The impressions and feedback from users after testing the App.
3. The obstacles and enablers to the App's use.
4. The expectations and needs of users for better use of the App.

The study's objectives include analyzing the usage behaviors, impressions, barriers, and needs of both young and older adults. It is a qualitative study based on non-participatory observations and semi-structured interviews with young and older participants who have used the App.

The App is based on impressionist artworks, a style known for evoking positive emotions, and aims to promote mental health by harnessing the emotional power of digital art and artificial intelligence.

ELIGIBILITY:
1. For adults of any age:

   1. Inclusion criteria:

      * Concordance of sex and gender.
      * No psychiatric or cognitive disorders.
      * Ability to understand spoken and written French.
      * Provide written consent to participate in the study.
   2. Exclusion criteria:

      * Non-binary.
      * Inability to provide informed consent to participate in the study.
      * Participation in a concurrent experimental clinical study to avoid interference with our study.
      * Inability to understand spoken and written French.
      * Having moderate to severe visual or auditory impairment.
2. Young adults:

   The inclusion criterion is being aged between 18 and 35 years.
3. Older adults:

The inclusion criterion is being aged 60 years or older.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Concordance of sex and gender
Enrollment: 30 (Estimated)
Dates: Start 2025-01-22 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Observation grid for behaviors and difficulties encountered | Day 1, during the use of the app, duration : 30 minutes
  Observation guide. Observation by a member of the research team will examine how participants use the App, in order to document usage behaviors and difficulties encountered.
Impressions and feedback | Day 1, right after the use of the app, duration : 30 minutes
  Semi-structured interview. The characteristics of these interviews are as follows:
  Format: The interviews are conducted with the participant and one or two members of the principal researcher's team.
  Interview guide: A structured guide is used to organize, standardize, and systematize the collection of information. This guide covers the following topics: impressions of the App (design, aesthetics, usability); participant's digital skills and abilities (integration and understanding of the tool); ease of interaction, enablers and barriers; impressions of AI in general; expectations, needs, and interests in such an App.
  Recording: With the participants' consent, the interviews are audio-recorded. The recording will be done using Audacity software, with the aim of producing a verbatim transcript for data analysis.
  Duration: 30 minutes.
Enablers and barriers | Day 1, right after the use of the app, duration : 30 minutes
  Semi-structured interview. The characteristics of these interviews are as follows:
  Format: The interviews are conducted with the participant and one or two members of the principal researcher's team.
  Interview guide: A structured guide is used to organize, standardize, and systematize the collection of information. This guide covers the following topics: impressions of the App (design, aesthetics, usability); participant's digital skills and abilities (integration and understanding of the tool); ease of interaction, enablers and barriers; impressions of AI in general; expectations, needs, and interests in such an App.
  Recording: With the participants' consent, the interviews are audio-recorded. The recording will be done using Audacity software, with the aim of producing a verbatim transcript for data analysis.
  Duration: 30 minutes.
Expectations and needs | Day 1, right after the use of the app, duration : 30 minutes
  Semi-structured interview. The characteristics of these interviews are as follows:
  Format: The interviews are conducted with the participant and one or two members of the principal researcher's team.
  Interview guide: A structured guide is used to organize, standardize, and systematize the collection of information. This guide covers the following topics: impressions of the App (design, aesthetics, usability); participant's digital skills and abilities (integration and understanding of the tool); ease of interaction, enablers and barriers; impressions of AI in general; expectations, needs, and interests in such an App.
  Recording: With the participants' consent, the interviews are audio-recorded. The recording will be done using Audacity software, with the aim of producing a verbatim transcript for data analysis.
  Duration: 30 minutes.

SECONDARY OUTCOMES:
Sociodemographics | Day 1
  A sociodemographic questionnaire is administered before using the App. This data is collected by a member of the principal researcher's (PR) team. It includes:
  Date of birth Sex and gender Ethnicity Native language Level of education Professional activity (past or current) or field of study Income level.
level of visual art knowledge | Day 1
  The Vienna Art Interest and Art Knowledge scale (VAIAK). The VAIAK is a psychometric scale developed to assess two main aspects related to art: personal interest in art and level of artistic knowledge. Due to the complexity of the scale and the number of questions, we will only use the part of the scale that evaluates interest in art. This part of the scale measures a person's interest and engagement with art. It includes aspects such as the frequency of museum visits, interest in different forms of art, and personal involvement in artistic activities. This section is divided into two subscales: the first asks, in 8 questions, to define the personal importance given to art and the enjoyment derived from these experiences on a 7-point scale ranging from "not at all" to "extremely." The second asks, in 4 questions, to define the frequency of interactions with art on a 7-point scale ranging from "less than once a year" to "once a week or more."
level of music knowledge | Day 1
  The Music Engagement Questionnaire (MusEQ). The MusEQ is used to explore the benefits of musical engagement in terms of cognitive and emotional regulation, active production, social connection, and physical exercise. This scale contains 32 questions that the participant answers using a 5-point Likert scale. These questions are divided into 6 subscales, which assess: 1) daily behavior related to music, 2) emotions, 3) practice, 4) consumption, 5) behavior, and 6) preferences. The scores for each subscale are calculated based on a combination of the responses.
Ecoanxiety level - Climate change | Day 1
  The Climate Change Anxiety Scale (CCAS): developed by Clayton & Karaszia, this climate change anxiety scale measures the emotional response to climate change through 22 items. It includes four subscales: cognitive and emotional impairment, functional impairment, personal experience of climate change, and behavioral engagement. Each item is rated on a 5-point Likert scale ranging from "Never" to "Almost always," scoring from 0 to 4 points for a total score between 0 and 88. The higher the score, the greater the level of eco-anxiety. A low score indicates relatively low anxiety related to climate change. The thresholds used in this project are: 0 to 22: low anxiety, 23 to 44: moderate anxiety, 45 to 66: high anxiety, and 67 to 88: very high anxiety.
Ecoanxiety level - Environmental issues | Day 1
  The Hogg Eco-Anxiety Scale (HEAS-13): developed by Hogg, this 13-item scale measures anxiety in response to environmental issues and the climate crisis, approaching eco-anxiety from an ecological perspective. Each item is rated on a 4-point Likert scale ranging from "Never" to "Almost every day," scoring from 0 to 3 points for a total score between 0 and 39. A low score indicates relatively low anxiety related to ecological issues. The thresholds used in this project are: 0 to 12: low anxiety, 13 to 25: moderate anxiety, and 26 to 39: high anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- CRIUGM, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided